CLINICAL TRIAL: NCT02056535
Title: Screening and Brief Intervention in the ED Among Mexican-origin Young Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Public Health Institute, California (Other)
Responsible Party: Principal Investigator, Cheryl Cherpitel, Senior Scientist, Public Health Institute, California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AA018119 (NIH)
Record Dates: First submitted 2013-06-04; First posted 2014-02-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2013-06

CONDITIONS: Problem Drinking; Alcohol Dependence
Keywords: Alcohol; SBIRT (Screening, Brief Intervention, Referral to Treatment)
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Screened Only (No Intervention): Screened only and met criteria for eligibility for study
- Screened and Assessed (No Intervention): Screened as eligible for the study and received baseline assessment
- Intervention (Active Comparator): Screened eligible, received baseline assessment and intervention
  Interventions: Behavioral: Brief Motivational Intervention

INTERVENTIONS:
Behavioral: Brief Motivational Intervention — A short discussion is held with patients identifying pros and cons of their drinking, readiness for change is assessed, and a brief prescription drawn for behavior change signed by the patient.
  Arms: Intervention

SUMMARY:
The aims of this study are to: 1) examine the effectiveness of Screening, Brief Intervention and Referral to Treatment (SBIRT) among Mexican-origin young adults (age 18-25), using a motivational intervention delivered by a Health Promotion Advocate, relative to standard care with and without assessment, on a reduction in heavy drinking and alcohol-related problems in the emergency department (ED) at the U.S.-Mexico border; and, 2) identify variables that are related to effectiveness of the intervention and that predict successful treatment outcome. Patients will be re-assessed by telephone at three and twelve months to evaluate outcomes.The specific hypotheses to be examined in this proposal are: 1) the motivational interview will lead to significantly greater reductions in the maximum number of drinks on an occasion and in Rapid Alcohol Problem Screen (RAPS4) score at the 12-month follow-up compared to standard care without assessment (those who screen positive but are not assessed) as well as compared to standard care with assessment; 2) the motivational interview will lead to significantly greater reductions in number of drinking days per week, average number of drinks per day, maximum number of drinks on an occasion, RAPS4 score, and number of negative consequences of drinking at 3-month and 12-month follow-up compared to standard care with assessment; 3) a positive breath alcohol concentration (BAC) at the time of the ED visit and/or self-reported drinking prior to the event resulting in the ED visit will be positively predictive of effectiveness of the intervention; 4) attributing a causal association of drinking and the reason for the ED visit will be positively associated with effectiveness of brief intervention; 5) readiness to change (and stage of change) will be positively associated with effectiveness of brief intervention; 6) risk taking/impulsivity and sensation seeking dispositions will be negatively associated with effectiveness of brief intervention.

DETAILED DESCRIPTION:
This is a randomized controlled brief intervention trial for dependent and at-risk drinking, among Mexican origin young adults (18-30) admitted to Texas Tech Health Sciences Center ER in El Paso, Texas, using Screening, Brief Intervention and Referral to Treatment (SBIRT) Patients are randomized into one of three groups: 1) screened only, 2) screened plus assessment, 3) screened plus assessment plus intervention with three-month outcome follow-up for the assessed and intervention groups and 12-month outcome follow-up for all three groups.

ELIGIBILITY:
Inclusion Criteria:

18-30 years old

1. Self-identify as Mexican-origin
2. Living in the El Paso area on the U.S. side
3. Screen positive for at-risk or dependent drinking (positive on one or more of the four RAPS4 items during the last year, or reports 15 or more drinks per week for males (8 or more for females), or reports 5 or more drinks on an occasion for males (4 or more for females)
4. Agree to be randomized to one of three groups
5. Can supply contact information on at least two individuals who will always know where they are
6. Not currently being treated for an alcohol problem

Exclusion Criteria:

* Does not meet inclusion criteria

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 698 (Actual)
Dates: Start 2010-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in the number of drinks per week and the number of drinks per drinking day | Baseline, 3 months & 12 months
  Change to less than 15 or more drinks per week for males (8 or more per week for females), and 5 or more drinks on occasion for males (4 or more for females)

SECONDARY OUTCOMES:
Change in Frequency of Drinking | Baseline, 3 months & 12 months
  Change in number of drinking days per week
Change in Alcohol-related problems | Baseline, 3 months &12 months
  Change in Rapid Alcohol Problem Screen score and Short Inventory of Problems related to drinking
Change in Quantity of Drinking | Baseline, 3 months & 12 months
  Change in average number of drinks per week; number of drinks per drinking day; and maximum number of drinks

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University Medical Sciences Center, ER, El Paso, Texas, United States

REFERENCES:
- [Derived] Cherpitel CJ, Ye Y, Bond J, Woolard R, Villalobos S, Bernstein J, Bernstein E, Ramos R. Brief Intervention in the Emergency Department Among Mexican-Origin Young Adults at the US-Mexico Border: Outcomes of a Randomized Controlled Clinical Trial Using Promotores. Alcohol Alcohol. 2016 Mar;51(2):154-63. doi: 10.1093/alcalc/agv084. Epub 2015 Aug 4. PMID 26243733